CLINICAL TRIAL: NCT03889912
Title: A Phase 1 Study of Pre-Operative Cemiplimab (REGN2810), Administered Intralesionally, for Patients With Cutaneous Squamous Cell Carcinoma (CSCC) or Basal Cell Carcinoma (BCC)
Brief Title: Intralesional Cemiplimab for Adult Patients With Cutaneous Squamous Cell Carcinoma or Basal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1787; 2024-511440-76-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2019-03-06; First posted 2019-03-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Basal Cell Carcinoma
Keywords: CSCC; BCC
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: Cohorts A, B, D and H will enroll sequentially (not randomized). Cohort C and I for BCC will enroll in parallel with, and independently of, Cohorts A, B, D and H for CSCC patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cemiplimab (Experimental): Three dose cohorts are planned and will follow a 3 + 3 dose-escalation design with cohort expansion. After completion of the above, three additional cohorts (A, B and C) of patients will be evaluated. Cohorts D, H and I may open after completion of Cohort B.
  Note: Cohort E through G will not be opened for participation.
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — Each patient will receive intralesional injections of cemiplimab every week (QW), or at less frequent dosing into the lesion at the assigned dose level for 3-12 weeks prior to scheduled surgery
  Other Names: REGN2810; Libtayo

SUMMARY:
This study is researching an experimental drug called cemiplimab. The study is focused on Cutaneous Squamous Cell Carcinoma (CSCC) and Basal Cell Carcinoma (BCC).

The aim of the study is to evaluate the safety and tolerability (how your body reacts to the drug) of cemiplimab (also known as REGN2810).

The first part of the study tested several different doses of cemiplimab given weekly for 12 weeks.

The study is also looking at several other research questions, including:

* What side effects may happen from taking the study drug
* To see effect of cemiplimab on the tumor
* How much study drug is in the blood at different times

ELIGIBILITY:
Key Inclusion Criteria

1. Dose Escalation: History of recurrent resectable CSCC or BCC (Cohort C and I only) that satisfies conditions as defined in the protocol
2. Patients must have measurable disease in the index lesion, defined as 1-2 cm in the longest diameter
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤1

Key Exclusion Criteria

1. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-mediated adverse events (imAEs)
2. Prior treatment with an agent that blocks the programmed cell death 1 (PD-1)/ programmed cell death 1 ligand (PD-L1) pathway.
3. Prior treatment with other systemic immune modulating agent as defined in the protocol
4. M1 or N1, N2 (a, b, or c), or N3 CSCC or BCC. Patients with history of metastatic CSCC (distant or nodal), or metastatic BCC (distant or nodal) are excluded unless the disease-free interval is at least 3 years
5. Concurrent malignancies, other than those with negligible risk of metastasis or death. Patients with hematologic malignancies, including chronic lymphocytic leukemia (CLL), are excluded.
6. Patients with a history of solid organ transplant
7. Has received a Coronavirus induced disease of 2019 (COVID-19) vaccination (initial series and booster) within 1 week of planned start of study medication

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Incidence, nature, and severity of dose limiting toxicities (DLTs) (if any) graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) v5 | From the first dose through day 28
  Dose levels 1-3
Incidence, nature, and severity of treatment-emergent adverse events (TEAEs) graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) v5 | From the first dose to 90 days after the last dose
  Dose levels 1-3
Incidence and severity of TEAEs graded according to the NCI CTCAE v5 | From the first dose up to 90 days after the last dose
The incidence and severity of injection site reactions (ISRs) | From the first dose to 90 days after the last dose

SECONDARY OUTCOMES:
Objective response rate (ORR) of index lesion | At baseline and at Week 13
  Determined by the investigator using the modified World Health Organization (WHO) criteria
Pathologic complete response rate (or end of treatment biopsies, for patients who decline surgery) in index lesion | At time of surgery
Major pathologic response rate (or end of treatment biopsies, for patients who decline surgery) in index lesion | At time of surgery
Cemiplimab concentration in serum over time | From the first dose up to 90 days after the last dose
Incidence of anti-drug antibody (ADA) titers for cemiplimab | Up to 90 days after last dose
Selection of the recommended dose of cemiplimab for further study based on clinical and pharmacokinetic (PK) observations | Up to 90 days after last dose
  The determination of the phase 2 recommended dose will be based primarily on clinical safety observations, according to the dose escalation scheme.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (18):
- United States (9):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - TCR Medical Corporation, San Diego, California
  - Dermatology Associates of the Palm Beaches, Delray Beach, Florida
  - MetroDerm, Atlanta, Georgia
  - Northeast Dermatology Associates, Beverly, Massachusetts
  - Rochester Dermatologic Surgery, P.C., Victor, New York
  - Duke Cancer Center, Durham, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
- Australia (4):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Netherlands (5):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - The Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, North Holland
  - University of Groningen, University Medical Centre Groningen, Groningen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/